CLINICAL TRIAL: NCT02762058
Title: Virtual Reality Mirror Therapy for Those With Acquired Brain Injury: A Clinical Pilot Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Guelph (Other)
Collaborators: Hamilton Health Sciences Corporation (Other); Natural Sciences and Engineering Research Council, Canada (Other)
Responsible Party: Principal Investigator, Laura MacNeil, Masters Student, University of Guelph
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1227
Record Dates: First submitted 2016-04-28; First posted 2016-05-04 (Estimated); Last update posted 2016-05-04 (Estimated); Status verified 2016-05

CONDITIONS: Acquired Brain Injury Including Stroke
Keywords: Acquired Brain Injury; Stroke Rehabilitation
MeSH Terms: conditions — Brain Injuries | interventions — Mirror Movement Therapy

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Experimental Group (Experimental): Patients receiving Virtual Reality Mirror Therapy
  Interventions: Device: Virtual Reality Mirror Therapy
- Control Group (Experimental): Patients receiving Traditional Mirror Therapy
  Interventions: Procedure: Traditional Mirror Therapy

INTERVENTIONS:
Device: Virtual Reality Mirror Therapy — Virtual Reality Mirror Therapy system using occulus rift as virtual headset and kinect as motion tracking sensor.
  Other Names: VMT; Occulus Rift; Microsoft Kinect
  Arms: Experimental Group
Procedure: Traditional Mirror Therapy — Traditional Mirror Therapy system consisting of a mirror in which patients view their healthy limb over the affected to trick brain during dual motion tasks. This therapy has been shown to improve upper extremity function in patients with acquired brain injury.
  Other Names: Mirror Therapy
  Arms: Control Group

SUMMARY:
The goal of this study is to investigate the effects of virtual reality based mirror therapy (VMT) on individuals with acquired brain injury when compared to a control group receiving traditional mirror therapy (TMT). This is a randomized controlled pilot study in which patients with hemiplegia will be assigned to VMT or TMT and the impact on upper extremity function will be observed.

DETAILED DESCRIPTION:
The investigators are currently running a mirror therapy pilot project in the Hamilton Health Sciences Rehabilitation Program. Mirror therapy has been successfully used with people that have injuries such as strokes or other types of brain injuries that affect movement on one side of their body. Mirror therapy involves placing a mirror over the affected limb and angling it to reflect the unaffected limb. This creates a visual illusion that moving the unaffected limb also results in movement in the affected limb. This is theorized to aid recovery of the motor system in the brain. Virtual Reality (VR) can also be used with people with strokes and brain injuries and many studies of VR have shown positive results. In this study, the investigators will combine VR and mirror therapy. The investigators have designed a special new system that uses VR headset to make it appear that both limbs are moving when only the unaffected limb is moving. The investigators are going to do this by having people complete virtual tasks wearing this specially programmed headset. The tasks are everyday activities that a person might perform using two hands. Ultimately, the investigators hope to determine whether there is any difference between VR mirror therapy and regular mirror therapy in improving upper limb function.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of stroke or brain injury, including ischemic or hemorrhagic strokes, confirmed by radio logical evidence and evidence suggesting injury primarily to one side and exhibited by hemiplegia
* their post injury time is between 2 weeks and 2 years
* patients are between the age of 16 and 65 years old

Exclusion Criteria:

* greater than stage 4 on the CMSA
* behavioral impairments that may prevent safe or consistent participation

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2016-06; Primary Completion 2019-06 (Estimated); Study Completion 2019-06 (Estimated)

PRIMARY OUTCOMES:
Upper Extremity Function | 6-weeks
  To measure subjects upper extremity function via assessment scores pre and post treatment.

SECONDARY OUTCOMES:
Upper Extremity Range of Motion | 6-weeks
  Arm position data recorded through the VR systems measured in millimeters.

OTHER OUTCOMES:
Mean Average Response Time | 6-weeks
  Mean average response time to complete tasks measured in seconds.

CONTACTS AND LOCATIONS:
Overall Officials: Hussein Abdullah, PhD, Principal Investigator — University of Guelph

IPD SHARING:
Plan to Share IPD: Undecided